CLINICAL TRIAL: NCT05308316
Title: Impact of Sugars on Tobacco Product Toxicity and Abuse Liability
Brief Title: Sugars in Cigarettes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2020LS236; R01DA051005 (NIH)
Record Dates: First submitted 2022-02-25; First posted 2022-04-04 (Actual); Results first posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Tobacco Use
MeSH Terms: conditions — Tobacco Use | interventions — Tobacco Products

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Impact of Sugar Content (Experimental): Participants will be asked to attend 4 laboratory sessions during which they will smoke their usual brand (UB) cigarettes and then one of three study cigarettes with low, medium and high levels of sugar in separate sessions, using a within-subject design with conditions counterbalanced determined by a Latin square. In each session, smokers will be asked to smoke a cigarette in a standardized manner (10 puffs,30 second interval between puffs) and 1 hour later, ad libitum. Each of the sessions will be separated by at least 48 hours but not more than 5 days.
  Interventions: Other: Cigarettes with added sucrose

INTERVENTIONS:
Other: Cigarettes with added sucrose — Winston brand cigarettes will be modified by adding sucrose to each cigarette at 2 levels so that the amount of total (originally present and added) sugar content in these cigarettes matches median and highest levels found in popular cigarette brands.

SUMMARY:
The aim of this study is to investigate the impact of sugar levels in cigarette tobacco on cigarette abuse liability and appeal. Participants will attend several clinic visits to smoke cigarettes with different levels of sugars and will complete multiple questionnaires to assess their experiences. Each of the sessions will be separated by at least 48 hours but not more than 5 days. The hypothesis is that the measures collected in this study will indicate lower abuse liability for cigarettes with lowest sugar content.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 21 years or older
* Smoking cigarettes that have been evaluated to have medium levels of sugar content
* No quit attempts in the past month nor intentions to quit smoking in the next month
* Participants are in good physical health (no unstable medical conditions) as determined by the licensed medical professional
* Participants are in stable, good mental health (e.g. not currently, within the past 6 months, experiencing unstable or untreated psychiatric diagnosis) as determined by the licensed medical professional
* Stable vitals sign measurements (systolic BP ≤ 160 and >90 mmHg, diastolic BP ≤ 100 and >50 mmHg and heart rate ≤105 and > 45 bpm) as determined by the licensed medical professional
* Participants must be able to read for comprehension or completion of study documents (confirmed during informed consent process)
* Participants have provided written informed consent to participate in the study.

Exclusion Criteria:

* Significant immune system disorders, respiratory diseases, kidney or liver diseases or any other medical disorders that may affect biomarker data as determined by the licensed medical professional
* Women who are pregnant or nursing or planning to become pregnant.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2026-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Irina Stepanov, PhD, Principal Investigator — University of Minnesota, Division of Environmental Health Sciences; Dorothy Hatsukami, Principal Investigator — Masonic Cancer Center Tobacco Research Programs
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants completed all three arms/sugar levels for the duration of the study.
Pre-assignment Details: Prior to being randomized to order of smoking study cigarettes all participants smoked their usual brand cigarettes. Each participant smoked all 3 versions of the study cigarettes (i.e., the 3 sugar levels). Participants were randomized to the order of smoking these different versions of cigarettes.
  Participants did not complete study due to withdrawal and physician decision.
Groups:
- Impact of Sugar Content: All Participants: After completing baseline assessment, participants will be asked to attend 3 laboratory sessions during which they will be asked to smoke one of three study cigarettes with low, medium and high levels of sugar in separate sessions using a within-subject design with conditions counterbalanced determined by a Latin square. In each session, smokers will be asked to smoke a cigarette in a standardized manner (10 puffs,30 second interval between puffs) and 1 hour later, ad libitum. Each of the sessions will be separated by at least 48 hours but not more than 5 days.
  Sucrose cigarettes: Winston brand cigarettes will be modified by adding a mixture of sucrose to each cigarette at 2 levels so that the amount of total (originally present and added) sugar content in these cigarettes matches median and highest levels found in popular brands analyzed
Period: Overall Study
Arm/Group | Impact of Sugar Content: All Participants
Started | 30
Usual Brand | 27
Low Sugar | 27
Medium Sugar | 27
High Sugar | 27
Completed | 27
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Impact of Sugar Content: All Participants
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.1 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 25
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Impact of Cigarette Sugar Content on Product Satisfaction.
Description: Product satisfaction will be measured using Modified Cigarette Evaluation Questionnaire (mCEQ). The mCEQ will involve 5 items rated on a 7-point Likert scale ranging from 1 "Not at all" to 7 "Extremely". A lower score would indicate less satisfaction, enjoyment smoking the assigned cigarette.
Time Frame: At each session, 2 hours post all puffs (assessed at all 4 sessions, each session was up to 4 hours, and all sessions took place between 2-3 weeks post enrollment, separated by 2-5 days)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Low Sugar Content; Medium Sugar Content; High Sugar Content: After completing baseline assessment, participants will be asked to attend 3 laboratory sessions during which they will be asked to smoke one of three study cigarettes with low, medium and high levels of sugar in separate sessions using a within-subject design with conditions counterbalanced determined by a Latin square. In each session, smokers will be asked to smoke a cigarette in a standardized manner (10 puffs,30 second interval between puffs) and 1 hour later, ad libitum. Each of the sessions will be separated by at least 48 hours but not more than 5 days.
  Sucrose cigarettes: Winston brand cigarettes will be modified by adding a mixture of sucrose to each cigarette at 2 levels so that the amount of total (originally present and added) sugar content in these cigarettes matches median and highest levels found in popular brands analyzed
- Usual Brand Cigarette: Prior to being randomized to order of smoking study cigarettes all participants smoked their usual brand cigarettes.
Arm/Group | Low Sugar Content | Medium Sugar Content | High Sugar Content | Usual Brand Cigarette
Number analyzed (Participants) | 25 | 25 | 25 | 25
units on a scale | 4.09 (1.85) | 3.89 (1.77) | 3.92 (1.87) | 4.39 (1.33)

2. Primary Outcome: Impact of Sugar Content on Behavioral Outcomes Using the Multiple Choice Procedure Task.
Description: Outcome measures for the Multiple Choice Procedure task are breakpoint (price at which participant switches from the study cigarette to money), elasticity (changes in consumption in response to changes in price); intensity (consumption at $0.00 price); Omax (maximum expenditure); and Pmax (price corresponding to Omax). Multiple Choice Procedure determines the price at which participants would switch from product to money, called the crossover point. Products with lower abuse liability tend to have a lower crossover point.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Dollars
Arm/Group | Low Sugar Content | Medium Sugar Content | High Sugar Content | Usual Brand Cigarette
Number analyzed (Participants) | 25 | 25 | 25 | 25
Dollars | 47.6 (123.64) | 27.20 (99.77) | 72.40 (147.8) | 113.8 (159.5)

3. Secondary Outcome: Other Subjective and Behavioral Measures: Effects/Liking
Description: Drug Effects/Liking Questionnaire is used to assess abuse liability of drugs and measures overall desirability of the product and intention to use in the future. Range from 0 - 100. A score of 0 being the weakest possible score, with 100 being the strongest score. Answers to questionnaire are averaged to calculate a composite score.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Low Sugar Content | Medium Sugar Content | High Sugar Content | Usual Brand Cigarette
Number analyzed (Participants) | 25 | 25 | 25 | 25
units on a scale | 47.85 (29.59) | 44.40 (27.70) | 47.33 (27.07) | 66.45 (23.40)

4. Secondary Outcome: Other Subjective and Behavioral Measures: Sensory Effect of Smoking
Description: Sensory Effect of Smoking Questionnaire (SESQ) uses a 7-point Likert scale ranging from 1 "Not at all" to 7 "Extremely", with a lower score indicating lower favorability, strength and effect of the cigarette on a participant. Five questions in this SESQ used for this study deal with the sensation of the strength of smoke impact on tongue, nose, mouth and throat, windpipe, and chest. Responses to each question were averaged to calculate final score. Total average minimum is one (lower effect) and total average maximum is seven (higher effect).
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Low Sugar Content | Medium Sugar Content | High Sugar Content | Usual Brand Cigarette
Number analyzed (Participants) | 25 | 25 | 25 | 25
units on a scale | 3.33 (0.78) | 3.16 (1.02) | 3.42 (1.22) | 3.29 (1.04)

5. Secondary Outcome: To Evaluate the Impact of Sugar Content on Smoking Intensity
Description: Measure the amount of nicotine levels in the spend filters during the controlled puffing pattern. Nicotine levels will be determined through LC/MS.
Time Frame: as for outcome 1
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Baseline to fourth session, up to 3 months
Groups:
- Impact of Sugar Content: Participants will be ask to attend 4 laboratory sessions during which they will be asked to smoke their usual brand (UB) cigarettes and then one of three study cigarettes with low, medium and high levels of sugar in separate sessions using a within-subject design with conditions counterbalanced determined by a Latin square. In each session, smokers will be asked to smoke a cigarette in a standardized manner (10 puffs,30 second interval between puffs) and 1 hour later, ad libitum. Each of the sessions will be separated by at least 48 hours but not more than 5 days.
  Sucrose cigarettes: Winston brand cigarettes will be modified by adding a mixture of sucrose to each cigarette at 2 levels so that the amount of total (originally present and added) sugar content in these cigarettes matches median and highest levels found in popular brands analyzed
Arm/Group | Impact of Sugar Content
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-01): https://cdn.clinicaltrials.gov/large-docs/16/NCT05308316/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/16/NCT05308316/ICF_001.pdf